CLINICAL TRIAL: NCT01257490
Title: Integrated Smoking Cessation Treatment for Low Income Community Corrections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Cropsey, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01CA141663 (NIH); R01CA141663 (NIH)
Record Dates: First submitted 2010-10-28; First posted 2010-12-09 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Counseling; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive counseling (Experimental): 4 sessions of intensive counseling plus bupropion
  Interventions: Behavioral: counseling vs. advice
- Brief Counseling (Active Comparator): Brief physician advice to quit plus bupropion
  Interventions: Behavioral: counseling vs. advice

INTERVENTIONS:
Behavioral: counseling vs. advice — 1 session of brief physician advice to quit smoking plus bupropion (12 weeks) compared to 4 sessions of intensive counseling plus bupropion (12 weeks)
  Other Names: counseling; wellbutrin; bupropion; zyban

SUMMARY:
This study recruited cigarette smokers under supervision in community corrections (e.g., probation, parole, drug courts, etc.) in the Birmingham, Alabama area. Smokers received 12 weeks of bupropion treatment and brief physician advice to quit smoking or 12 weeks of bupropion treatment and 4 sessions of intensive counseling around smoking cessation. The study was stratified on race such that equal proportions of African Americans and Caucasians were enrolled in the two study groups. It was hypothesized that smokers receiving intensive counseling will have higher quit rates compared to smokers receiving brief advice to quit.

ELIGIBILITY:
Inclusion Criteria:

* At least 19 years or older
* Enrolled in criminal justice community supervision (e.g., probation, parole, drug court, community corrections, etc)
* Smoking at least 5 cpd for the past year
* Maintained in an unrestricted environment (e.g., not currently in a correctional facility or treatment facility) living in the Birmingham Area and surrounding communities

Exclusion Criteria:

* Pregnant or nursing (all women in this study will be required to use an acceptable form of contraception throughout the administration of the medication)
* Known sensitivity to Zyban or Wellbutrin
* History of seizures
* Current or prior anorexia or bulimia
* Abrupt withdrawal from alcohol or benzodiazepines
* Moderate to severe kidney problems
* Moderate liver problems
* Cognitive impairment such that they cannot provide informed consent

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2009-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
smoking cessation | 3 months
smoking cessation | 6 Month
smoking cessation | 9 Month
smoking cessation | 12 Month

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Cropsey, Psy.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Substance Abuse, Birmingham, Alabama, United States